CLINICAL TRIAL: NCT00395876
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study of Tenecteplase for Restoration of Function in Dysfunctional Central Venous Catheters
Brief Title: A Study of Tenecteplase for Restoration of Function in Dysfunctional Central Venous Catheters
Acronym: TROPICS 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Clinical Trials Posting Group, Genentech, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N3698g
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Results first posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-07

CONDITIONS: Dysfunctional Central Venous Access Catheters
Keywords: TNKase; CVA; CVAD; Central venous access catheter; CVA catheter
MeSH Terms: interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo + Tenecteplase + Tenecteplase (PTT) (Placebo Comparator)
  Interventions: Drug: placebo; Drug: tenecteplase
- Tenecteplase + Tenecteplase + Placebo (TTP) (Experimental)
  Interventions: Drug: placebo; Drug: tenecteplase

INTERVENTIONS:
Drug: placebo — 2 mL of placebo instilled into lumen of dysfunctional CVC. Patients weighing ≥ 30 kg received 2-mL instillations of study drug (i.e., 2 mg of placebo). Patients weighing < 30 kg received instillations of study drug equal to 110% of the internal lumen volume of the dysfunctional CVC. This dose was rounded to the nearest 0.1 mL and should not have exceeded 2 mL (2 mg).
Drug: tenecteplase — 2 mL of reconstituted lyophilized tenecteplase instilled into lumen of dysfunctional CVC. Patients weighing ≥ 30 kg received 2-mL instillations of study drug (i.e., 2 mg of tenecteplase). Patients weighing < 30 kg received instillations of study drug equal to 110% of the internal lumen volume of the dysfunctional CVC. This dose was rounded to the nearest 0.1 mL and should not have exceeded 2 mL (2 mg).

SUMMARY:
This was a Phase III, randomized, double-blind, placebo-controlled study that was conducted at 24 centers in the United States and Canada. 100 adult and pediatric patients with dysfunctional central venous catheters (CVCs) were randomly assigned in a 1:1 ratio to receive an initial dose of either placebo (Arm A) or tenecteplase (Arm B).

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable, in the opinion of the investigator
* CVC occlusion
* Able to have fluids infused at the volume necessary to instill study drug into the CVC

Exclusion Criteria:

* Able to have 3 mL of blood (patients weighing ≥ 10 kg) or 1 mL of blood (patients weighing < 10 kg) withdrawn from the selected study CVC following patient repositioning
* Selected study CVC inserted < 2 days prior to treatment
* Selected study CVC known to be dysfunctional for > 7 days
* Selected study CVC implanted specifically for hemodialysis (HD)
* Use of a power injector on the selected study CVC during the study
* Evidence of mechanical, non-thrombotic occlusion of the selected study CVC (e.g., kink in the catheter or suture constricting the catheter)
* Previously treated in this study or any tenecteplase catheter clearance trial
* Use of any investigational drug or therapy within 28 days prior to treatment
* Use of a fibrinolytic agent (e.g., alteplase, tenecteplase, reteplase, or urokinase) within 24 hours prior to treatment
* Known to be pregnant or breastfeeding at screening
* CVC with known or suspected infection
* History of any intracranial hemorrhage, aneurysm, or arteriovenous malformation
* Use of heparin (unfractionated or low molecular weight) within 24 hours prior to treatment, except for use of intermittent or low-dose, continuous infusion of heparin to maintain catheter or vessel patency
* Use of warfarin within 7 days prior to treatment, except for low-dose warfarin used for prophylaxis
* Initiation of or increase in dose of Plavix® (clopidogrel bisulfate) within 7 days prior to treatment
* At high risk for bleeding events or embolic complications (i.e., recent pulmonary embolus, deep vein thrombosis, endarterectomy, or clinically significant right-to-left shunt) in the opinion of the investigator, or with known condition for which bleeding constitutes a significant hazard
* Known hypersensitivity to tenecteplase or any component of the formulation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-11; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Levine, M.D., Study Director

REFERENCES:
- [Derived] Gabrail N, Sandler E, Charu V, Anas N, Lim E, Blaney M, Ashby M, Gillespie BS, Begelman SM. TROPICS 1: a phase III, randomized, double-blind, placebo-controlled study of tenecteplase for restoration of function in dysfunctional central venous catheters. J Vasc Interv Radiol. 2010 Dec;21(12):1852-8. doi: 10.1016/j.jvir.2010.09.002. PMID 21111365

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three patients were randomized but not treated, therefore the modified intent to treat (MITT) analysis population was 97.
Groups:
- Placebo + Tenecteplase + Tenecteplase (PTT): Initial dose: 2 mL of placebo instilled into lumen of dysfunctional central venous cathether (CVC).
  If CVC function was not restored, patient received second dose: 2 mL of reconstituted lyophilized tenecteplase instilled into lumen of dysfunctional CVC.
  If CVC function was not restored, patient received third dose: 2 mL of reconstituted lyophilized tenecteplase instilled into lumen of dysfunctional CVC.
  Restoration of CVC function was defined as the successful withdrawal of at least 3 mL of blood or fluid and infusion of 5 mL of normal saline in patients weighing ≥ 10 kg, and withdrawal of at least 1 mL of blood or fluid and infusion of 3 mL of normal saline in patients weighing < 10 kg.
- Tenecteplase + Tenecteplase + Placebo (TTP): Initial dose: 2 mL of reconstituted lyophilized tenecteplase instilled into lumen of dysfunctional CVC.
  If CVC function not restored, patient received second dose: 2 mL of reconstituted lyophilized tenecteplase instilled into lumen of dysfunctional CVC.
  If CVC function not restored, patient received third dose: 2 mL of placebo instilled into lumen of dysfunctional CVC.
  Restoration of CVC function was defined as the successful withdrawal of at least 3 mL of blood or fluid and infusion of 5 mL of normal saline in patients weighing ≥ 10 kg, and withdrawal of at least 1 mL of blood or fluid and infusion of 3 mL of normal saline in patients weighing < 10 kg.
Period: Overall Study
Arm/Group | Placebo + Tenecteplase + Tenecteplase (PTT) | Tenecteplase + Tenecteplase + Placebo (TTP)
Started | 50 | 50
Completed | 47 | 50
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Tenecteplase + Tenecteplase (PTT) | Tenecteplase + Tenecteplase + Placebo (TTP) | Total
Number analyzed (Participants) | 47 | 50 | 97
Age, Customized [Number; unit: participants]
  < 2 years | 1 | 3 | 4
  ≥ 2 to < 17 years | 14 | 16 | 30
  ≥ 17 to < 65 years | 17 | 20 | 37
  ≥ 65 years | 15 | 11 | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 42.2 (28.3) | 37.1 (26.6) | 39.6 (27.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 26 | 57
  Male | 16 | 24 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Had Restoration of Central Venous Catheter (CVC) Function Following a Single Administration of Study Drug
Description: Restoration of CVC function was defined as successful withdrawal of at least 3 mL of blood or fluid and infusion of 5 mL of normal saline in patients weighing ≥ 10 kg, and withdrawal of at least 1 mL of blood or fluid and infusion of 3 mL of normal saline in patients weighing < 10 kg.
Time Frame: 120 minutes after first dose
Population: Modified intent to treat (MITT) population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Tenecteplase + Tenecteplase (PTT) | Tenecteplase + Tenecteplase + Placebo (TTP)
Number analyzed (Participants) | 47 | 50
percentage of participants | 23.4 | 60.0
Statistical Analysis 1: Comparison: Placebo + Tenecteplase + Tenecteplase (PTT) vs Tenecteplase + Tenecteplase + Placebo (TTP); Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel — Stratified by baseline weight (< 30 kg, ≥ 30 kg); Mean Difference (Final Values) = 36.6, 95% CI [18.4 to 54.8]

2. Secondary Outcome: Percentage of Patients Who Had Restoration of CVC Function Following a Single Administration of Study Drug
Description: as for outcome 1
Time Frame: 15 minutes after first dose
Population: Modified intent to treat (MITT) population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Tenecteplase + Tenecteplase (PTT) | Tenecteplase + Tenecteplase + Placebo (TTP)
Number analyzed (Participants) | 47 | 50
percentage of participants | 10.6 | 22.0
Statistical Analysis 1: Comparison: Placebo + Tenecteplase + Tenecteplase (PTT) vs Tenecteplase + Tenecteplase + Placebo (TTP); Test type: Superiority or Other; p = 0.1385, Cochran-Mantel-Haenszel — Stratified by baseline weight (< 30 kg, ≥ 30 kg); Mean Difference (Final Values) = 11.4, 95% CI [-3.1 to 25.8]

3. Secondary Outcome: Percentage of Patients Who Had Restoration of CVC Function Following a Single Administration of Study Drug
Description: as for outcome 1
Time Frame: 30 minutes after first dose
Population: Modified intent to treat (MITT) population
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo + Tenecteplase + Tenecteplase (PTT) | Tenecteplase + Tenecteplase + Placebo (TTP)
Number analyzed (Participants) | 47 | 50
Percentage of patients | 19.1 | 44.0
Statistical Analysis 1: Comparison: Placebo + Tenecteplase + Tenecteplase (PTT) vs Tenecteplase + Tenecteplase + Placebo (TTP); Test type: Superiority or Other; p = 0.0093, Cochran-Mantel-Haenszel — Stratified by baseline weight (< 30 kg, ≥ 30 kg); Mean Difference (Final Values) = 24.9, 95% CI [7.1 to 42.6]

4. Secondary Outcome: Percentage of Patients Who Had Restoration of CVC Function Following a Second Administration of Study Drug
Description: as for outcome 1
Time Frame: 15 minutes after second dose
Population: Modified intent to treat (MITT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Tenecteplase + Tenecteplase (PTT) | Tenecteplase + Tenecteplase + Placebo (TTP)
Number analyzed (Participants) | 47 | 50
percentage of participants | 42.6 [28.4 to 56.7] | 70.0 [57.3 to 82.7]

5. Secondary Outcome: Percentage of Patients Who Had Restoration of CVC Function Following a Second Administration of Study Drug
Description: as for outcome 1
Time Frame: 30 minutes after second dose
Population: Modified intent to treat (MITT) population
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Placebo + Tenecteplase + Tenecteplase (PTT) | Tenecteplase + Tenecteplase + Placebo (TTP)
Number analyzed (Participants) | 47 | 50
Percentage of patients | 63.8 [50.1 to 77.6] | 82.0 [71.4 to 92.6]

6. Secondary Outcome: Percentage of Patients Who Had Restoration of CVC Function Following a Second Administration of Study Drug
Description: as for outcome 1
Time Frame: 120 minutes after second dose
Population: Modified intent to treat (MITT) population
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Placebo + Tenecteplase + Tenecteplase (PTT) | Tenecteplase + Tenecteplase + Placebo (TTP)
Number analyzed (Participants) | 47 | 50
Percentage of patients | 72.3 [59.6 to 85.1] | 88.0 [79.0 to 97.0]

7. Secondary Outcome: Percentage of Patients Who Had Restoration of CVC Function Following a Third Administration of Study Drug
Description: as for outcome 1
Time Frame: 15 minutes after third dose
Population: Modified intent to treat (MITT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Tenecteplase + Tenecteplase (PTT) | Tenecteplase + Tenecteplase + Placebo (TTP)
Number analyzed (Participants) | 47 | 50
percentage of participants | 83.0 [72.2 to 93.7] | 88.0 [79.0 to 97.0]

8. Secondary Outcome: Percentage of Patients Who Had Restoration of CVC Function Following a Third Administration of Study Drug
Description: as for outcome 1
Time Frame: 30 minutes after third dose
Population: Modified intent to treat (MITT) population
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Placebo + Tenecteplase + Tenecteplase (PTT) | Tenecteplase + Tenecteplase + Placebo (TTP)
Number analyzed (Participants) | 47 | 50
Percentage of patients | 85.1 [74.9 to 95.3] | 88.0 [79.0 to 97.0]

9. Secondary Outcome: Percentage of Patients Who Had Restoration of CVC Function Following a Third Administration of Study Drug
Description: as for outcome 1
Time Frame: 120 minutes after third dose
Population: Modified intent to treat (MITT) population
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Placebo + Tenecteplase + Tenecteplase (PTT) | Tenecteplase + Tenecteplase + Placebo (TTP)
Number analyzed (Participants) | 47 | 50
Percentage of patients | 85.1 [74.9 to 95.3] | 88.0 [79.0 to 97.0]

10. Secondary Outcome: Percentage of Patients Who Had Restoration of CVC Function Following Administration of One or Two Doses of Tenecteplase
Description: Restoration of CVC function was defined as the successful withdrawal of at least 3 mL of blood or fluid and infusion of 5 mL of normal saline in patients weighing ≥ 10 kg, and withdrawal of at least 1 mL of blood or fluid and infusion of 3 mL of normal saline in patients weighing < 10 kg.
Time Frame: Up to 120 minutes post-treatment
Population: Modified intent to treat (MITT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Tenecteplase + Tenecteplase (PTT) | Tenecteplase + Tenecteplase + Placebo (TTP)
Number analyzed (Participants) | 47 | 50
percentage of participants
  Through first tenecteplase instillation | 72.3 [59.6 to 85.1] | 60.0 [46.4 to 73.6]
  Through second tenecteplase instillation | 85.1 [74.9 to 95.3] | 88.0 [79.0 to 97.0]

11. Secondary Outcome: Percentage of Patients Who Had Restoration of CVC Function at Any Time During the Study and Who Maintained Catheter Patency the Next Time the Catheter Was Assessed, up to 7 Days Following the Last Dose of Tenecteplase
Description: as for outcome 10
Time Frame: Up to 7 days post-treatment
Population: Number of patients (from MITT population) with restored CVC function during the treatment period
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Placebo + Tenecteplase + Tenecteplase (PTT) | Tenecteplase + Tenecteplase + Placebo (TTP)
Number analyzed (Participants) | 27 | 29
Percentage of patients | 81.5 [66.8 to 96.1] | 79.3 [64.6 to 94.1]

ADVERSE EVENTS:
Description: Modified intent to treat (MITT) population.
  Note: The incidence of each AE/SAE is reported as the number of participants experiencing the event, not the number of occurrences for each AE/SAE.
Arm/Group | Placebo + Tenecteplase + Tenecteplase (PTT) | Tenecteplase + Tenecteplase + Placebo (TTP)
Serious Adverse Events (participants affected / at risk) | 1/47 | 2/50
Other Adverse Events (participants affected / at risk) | 6/47 | 14/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Tenecteplase + Tenecteplase (PTT) (N=47) | Tenecteplase + Tenecteplase + Placebo (TTP) (N=50)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 1 | 0
Venous Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Tenecteplase + Tenecteplase (PTT) (N=47) | Tenecteplase + Tenecteplase + Placebo (TTP) (N=50)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdonimal Pain (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Catheter Site Pain (General disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Axillary Pain (General disorders) | 0 | 1
Catheter Site Oedema (General disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Central Line Infection (Infections and infestations) | 0 | 1
Escherichia Sepsis (Infections and infestations) | 0 | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 1
Platelet Count Decreased (Investigations) | 0 | 1
Weight Decreased (Investigations) | 0 | 1
Hypertriglycerideaemia (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Burning Sensation (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Glycosuria (Renal and urinary disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Haematoma (Vascular disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.